CLINICAL TRIAL: NCT03633968
Title: Assessment of the Effect of the Antrostomy Size in Graftless Lateral Maxillary Sinus Floor Elevation Using AMBE (Antral Membrane Balloon Elevation) With Simultaneous Implant Placement
Brief Title: Graftless Lateral Maxillary Sinus Lift Balloon by Different Antrostomy Sizes With Simultaneous Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ahmed mohammed khalil aldahouk (Other)
Responsible Party: Sponsor-Investigator, ahmed mohammed khalil aldahouk, Principal Investigator(doctor), Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: maxillary sinus augmentation
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Atrophy of Edentulous Maxillary Alveolar Ridge
Keywords: sinus augmentation,lifting

STUDY DESIGN:
Intervention Model Description: assessment of the effect of the antrostomy size in graftless lateral maxillary sinus floor elevation using AMBE (antral membrane balloon elevation) with simultaneous implant placement
Who Masked: Participant
Masking Description: assessment of the effect of the antrostomy size in graftless lateral maxillary sinus floor elevation using AMBE (antral membrane balloon elevation) with simultaneous implant placement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maxillary sinus lift small antrostomy (Active Comparator): local anaesthesia will be given flap will be reflected to expose sinus lateral wall. round diamond bur will be used to make small antrostomy and expose schneiderian membrane.
  maxillary sinus lift by using antral membrane balloon elevation without using graft material with simultaneous implant placement
  Interventions: Procedure: maxillary sinus lift
- maxillary sinus lift large antrostomy (Active Comparator): local anaesthesia will be given flap will be reflected to expose sinus lateral wall round diamond bur will be used to make large antrostomy and expose schneiderian membrane.
  maxillary sinus lift by using antral membrane balloon elevation without using graft material with simultaneous implant placement
  Interventions: Procedure: maxillary sinus lift

INTERVENTIONS:
Procedure: maxillary sinus lift — maxillary sinus floor elevation by using balloon through either small or large antrostomy without using graft material with simultaneous implant placement
  Other Names: implant placement

SUMMARY:
two groups undergo for graftless sinus lift using AMBE (antral membrane balloon elevation) through different antrostomy size with simultaneous implant placement

DETAILED DESCRIPTION:
control group undergoes for graftless sinus lift using AMBE through large antrostomy with simultaneous implant placement. While, study group undergo for graftless sinus lift using AMBE through small antrostomy with simultaneous implant placement. the aim of the study is assessment the effect of antrostomy size on bone formation in graftless sinus lift with simultaneous implant placement.

CBCT will be done before and after the surgery and after 6 months to assess of amount bone gain in mm.

implant stability after 6 months will be determined by using Osstell. Primary outcome: amount of bone gain which will be measured by using linear measurement from CBCT.

secondary outcome: stability of implant by using osstell

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atrophic maxilla and pneumatization of maxillary sinus with residual bone height from 3-6mm.
2. Both sexes
3. No intraoral soft and hard tissue pathology,
4. No systemic condition that contraindicate implant placement

Exclusion Criteria:

1. Sinus pathology.
2. Heavy smokers more than 20 cigarettes per day.
3. Patients with systemic disease that may affect normal healing.
4. Psychiatric problems.
5. Disorders to implant are related to history of radiation therapy to head and neck neoplasia or bone augmentation to implant site

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
amount of bone formation | after 6 months
  measurement of amount of bone gained by using CBCT

SECONDARY OUTCOMES:
implant stability | after 6 months
  measurement of implant stability by using osstell

CONTACTS AND LOCATIONS:
Overall Officials: ahmed a dahouk, bsd, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Al-Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
web sites and journals

REFERENCES:
- [Background] Stern A, Green J. Sinus lift procedures: an overview of current techniques. Dent Clin North Am. 2012 Jan;56(1):219-33, x. doi: 10.1016/j.cden.2011.09.003. PMID 22117952
- [Background] Summers RB. The osteotome technique: Part 3--Less invasive methods of elevating the sinus floor. Compendium. 1994 Jun;15(6):698, 700, 702-4 passim; quiz 710. PMID 7994726
- [Background] Soltan M, Smiler DG. Antral membrane balloon elevation. J Oral Implantol. 2005;31(2):85-90. doi: 10.1563/0-773.1. PMID 15871527
- [Background] Esposito M, Grusovin MG, Rees J, Karasoulos D, Felice P, Alissa R, Worthington H, Coulthard P. Effectiveness of sinus lift procedures for dental implant rehabilitation: a Cochrane systematic review. Eur J Oral Implantol. 2010 Spring;3(1):7-26. PMID 20467595
- [Background] Watanabe T, Nakagawa E, Saito K, Ohshima H. Differences in Healing Patterns of the Bone-Implant Interface between Immediately and Delayed-Placed Titanium Implants in Mouse Maxillae. Clin Implant Dent Relat Res. 2016 Feb;18(1):146-60. doi: 10.1111/cid.12280. Epub 2015 Apr 15. PMID 25872947
- [Background] Avila-Ortiz G, Wang HL, Galindo-Moreno P, Misch CE, Rudek I, Neiva R. Influence of lateral window dimensions on vital bone formation following maxillary sinus augmentation. Int J Oral Maxillofac Implants. 2012 Sep-Oct;27(5):1230-8. PMID 23057039
- [Background] Testori T, Weinstein RL, Taschieri S, Del Fabbro M. Risk factor analysis following maxillary sinus augmentation: a retrospective multicenter study. Int J Oral Maxillofac Implants. 2012 Sep-Oct;27(5):1170-6. PMID 23057031
- [Background] Hatziotis JC, Papanayotou PH, Trigonidis G. Benign mesenchymoma of the tongue: report of case. J Oral Surg. 1972 Jan;30(1):45-6. No abstract available. PMID 4500328
- [Background] Barone A, Santini S, Marconcini S, Giacomelli L, Gherlone E, Covani U. Osteotomy and membrane elevation during the maxillary sinus augmentation procedure. A comparative study: piezoelectric device vs. conventional rotative instruments. Clin Oral Implants Res. 2008 May;19(5):511-5. doi: 10.1111/j.1600-0501.2007.01498.x. Epub 2008 Mar 26. PMID 18371101